CLINICAL TRIAL: NCT01582139
Title: Feasibility Study of Closed Loop Control in Type 1 Diabetes Using Heart Rate Monitoring as an Exercise Marker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); DexCom, Inc. (Industry); Insulet Corporation (Industry); Abbott Diabetes Care (Industry)
Responsible Party: Principal Investigator, Marc Breton, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15970; 5R21DK085641 (NIH)
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas Project; AP Platform; Insulin Pump; Continuous Glucose Monitor; Closed-Loop Control; Control-to-Range
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Condition: (Heart-Rate Informed SSM+HMM) (Experimental): An experimental condition involving an exercise session where the Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) is informed about heart rate
  Interventions: Device: Heart rate informed SSM+HMM
- Control Condition (SSM+HMM) (No Intervention): A control condition involving an exercise session where the Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) is not informed about heart rate.

INTERVENTIONS:
Device: Heart rate informed SSM+HMM — The Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) of the Closed Loop is informed about heart rate during exercise. The goal is to demonstrate the feasibility of a modular insulin management system based on continuous glucose monitoring that additionally employs heart rate information to reduce exercise-related hypoglycemic episodes.
  Arms: Experimental Condition: (Heart-Rate Informed SSM+HMM)

SUMMARY:
The purpose of this study is to see if the Artificial Pancreas Platform (AP Platform = Cell Phone + Closed Loop Control) can successfully control blood sugar in people with type 1 diabetes mellitus on insulin pump therapy in a hospital setting. Investigators will also be studying to see if information about heart rate can help the AP Platform reduce hypoglycemia related to exercise.

DETAILED DESCRIPTION:
The combination of the Control to Range system and the cell phone is called the "Artificial Pancreas (AP) Platform". The purpose of this study is to see if this investigational technology can help control blood sugar in people with type 1 diabetes mellitus on insulin pump therapy can be successfully used and supervised in a hospital setting. This study is also being done to see if giving information about heart rate to the Closed-to-Range System can reduce hypoglycemia as it relates to exercise. Subjects will exercise on an exercise bike in the clinical research unit. During one exercise testing session, the Closed-to-Range System will receive information about your heart rate (Experimental Condition). During the other exercise testing session, the Control to Range System will not receive information about your heart rate (Control Condition). This part of the study is being done to see whether heart rate information helps the Closed-to-Range System reduce the occurrences of exercise-related hypoglycemia.

The Closed-to-Range system has two parts (modules) that can work together or separately.

A. The Safety Supervision Module (SSM) helps to prevent low blood sugars. It can reduce the amount of basal insulin that the pump is delivering and alert you if carbohydrates are needed to help prevent a low blood sugar. This module will be active at all times during the operation of the Closed-to-Range System.

B. The Hyperglycemia Mitigation Module (HMM) helps to prevent high blood sugars. It can instruct the insulin pump to deliver small boluses to help prevent high blood sugar. It can also help warn you of a possible pump problem if the blood sugar level is not responding to the insulin as it should.

The Closed-to-Range System works with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range (80-180 mg/dL) during the day and help avoid hypoglycemia during the night.

ELIGIBILITY:
Inclusion Criteria

1. ≥21 and <65 years old with clinical diagnosis of Type 1 Diabetes Mellitus for at least 1 year.
2. Criteria for documented hyperglycemia (at least 1 criterion must be met):

   1. Fasting glucose ≥126 mg/dL - confirmed
   2. Two-hour Oral Glucose Tolerance Test (OGTT) glucose ≥200 mg/dL - confirmed
   3. HbA1c ≥6.5% documented - confirmed
   4. Random glucose ≥200 mg/dL with symptoms
3. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes.

   Criteria for requiring insulin at diagnosis (at least 1 criterion must be met):
   1. Participant required insulin at diagnosis and continually thereafter
   2. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
   3. Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes (LADA) in adults and did require insulin eventually and used continually.

      Criteria for Type 1 Diabetes Mellitus (at least 1 criterion must be met)
   4. Documented low or absent C-peptide level.
   5. Documented presence of Islet Cell Cytoplasmic Autoantibodies (ICA) or Glutamic Acid Decarboxylase (GAD65) antibodies.
4. Use of an insulin pump to treat his/her diabetes for at least 6 months
5. Actively using a bolus calculator with the current insulin pump with pre-defined parameters for carbohydrate (CHO) ratio, insulin sensitivity factor (ISF), and target glucose
6. HbA1c between 5.0% and 10.5% as measured with DCA2000 or equivalent device
7. Not currently known to be pregnant, breast feeding, or intending to become pregnant (females)
8. Demonstration of proper mental status and cognition for the study.
9. Willingness to avoid consumption of acetaminophen-containing products during the study interventions involving continuous glucose monitor use.
10. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study.

Exclusion Criteria

1. Clinical diagnosis of Type 2 Diabetes Mellitus
2. Diabetic ketoacidosis within the 6 months prior to enrollment
3. Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment
4. Pregnancy, breast feeding, or intention of becoming pregnant
5. Uncontrolled arterial hypertension (diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg)
6. Hematocrit <36% (females); <38% (males)
7. Uncontrolled thyroid disease or thyroid replacement as determined by a thyroid-stimulating hormone (TSH) out of the UVa reference range.
8. Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase >2 times the upper limit of normal
9. Impaired renal function measured as creatinine >1.5 mg/dL
10. Conditions which may increase the risk of hypoglycemia such as known coronary artery disease (e.g. history of myocardial infarction, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, or positive stress test or catheterization with coronary blockages >50%), congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, adrenal insufficiency, neurologic disease or atrial fibrillation
11. Additional conditions which may inhibit the ability to perform exercise on a stationary bike (e.g. injury to or immobility of limbs, neuromuscular disease, exercise-induced asthma requiring inhaler use within the last 12 months or clinically impaired pulmonary function)
12. Use of a medication that significantly lowers heart rate (beta blockers, reserpine, guanethidine, methyldopa, clonidine, cimetidine, digitalis, calcium channel blockers, amiodarone, antiarrythmic drugs, or lithium)
13. History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans
14. Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the continuous glucose monitor (CGM) (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants)
15. Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for the study admissions.
16. Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment, uncontrolled anxiety or panic disorder)
17. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
18. Current or recent alcohol or drug abuse by patient history
19. Medical conditions that would make operating a CGM, cell phone or insulin pump difficult (e.g. blindness, severe arthritis, immobility)
20. Any skin condition that prevents sensor or pump placement on the abdomen or arm (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis)
21. Known microvascular (diabetic) complications (other than diabetic non-proliferative retinopathy), such as history of laser coagulation, proliferative diabetic retinopathy, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment
22. Active gastroparesis requiring current medical therapy
23. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
24. Known bleeding diathesis or dyscrasia
25. Known allergy to medical adhesives, components of the insulin pump insertion set or continuous glucose monitor sensor
26. Anticoagulant therapy other than aspirin
27. Oral steroids
28. Active enrollment in another clinical trial
29. Unwillingness to avoid acetaminophen while the continuous glucose monitor is in use.
30. Unwillingness to withhold dietary supplements two weeks prior to admission and for the duration of the study participation.
31. Subjects with basal rates less than 0.05.

Restrictions on use of other drugs or treatments

1. Pramlintide, liraglutide and exenatide will be held for the duration of the study intervention.
2. Oral steroids are excluded
3. Anticoagulant therapy other than aspirin is excluded
4. Acetaminophen will not be allowed while the continuous glucose monitor is in use
5. Dietary supplements will be withheld two weeks prior to admission and for the duration of study participation
6. Beta blockers, reserpine, guanethidine, methyldopa, clonidine, cimetidine, digitalis, calcium channel blockers, amiodarone, antiarrythmic drugs, and lithium are excluded

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Breton, Ph.D., Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Breton MD, Brown SA, Karvetski CH, Kollar L, Topchyan KA, Anderson SM, Kovatchev BP. Adding heart rate signal to a control-to-range artificial pancreas system improves the protection against hypoglycemia during exercise in type 1 diabetes. Diabetes Technol Ther. 2014 Aug;16(8):506-11. doi: 10.1089/dia.2013.0333. Epub 2014 Apr 4. PMID 24702135

RESULTS

PARTICIPANT FLOW:
Groups:
- Control First, Then Experimental; Experimental First, Then Control: Control, SSM+HMM: A control condition involving an exercise session where the Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) is not informed about heart rate.
  Experimental, Heart-Rate Informed SSM: An experimental condition involving an exercise session where the Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) is informed about heart rate
Period: Overall Study
Arm/Group | Control First, Then Experimental | Experimental First, Then Control
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control First, Then Experimental | Experimental First, Then Control | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemic Events
Description: Plasma glucose based number of hypoglycemic events, defined as consecutive plasma readings below 70mg/dl to measure the capacity of the system to protect patients against the risk of hypoglycemia. Two events separated by only one Yellow Springs Instrument (YSI) value over 70 are considered to form a single event.
Time Frame: 26 hours (x2 admissions)
Population: Twelve subjects completed the study. The first two subjects were excluded from the analysis because of protocol violations during the exercise session (the intensity chosen was very high: rating of perceived exertion of 9 out of 10 instead of rating of perceived exertion of 9 out of 20). Results from the 10 remaining subjects are presented below.
Measure: Number; unit: hypoglycemic events
Groups:
- Experimental: Heart-Rate Informed SSM+HMM: An experimental condition involving an exercise session where the Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) is informed about heart rate
  Heart rate informed SSM+HMM: The Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) of the Closed Loop is informed about heart rate during exercise. The goal is to demonstrate the feasibility of a modular insulin management system based on continuous glucose monitoring that additionally employs heart rate information to reduce exercise-related hypoglycemic episodes.
- Control: SSM+HMM: A control condition involving an exercise session where the Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) is not informed about heart rate.
Arm/Group | Experimental: Heart-Rate Informed SSM+HMM | Control: SSM+HMM
Number analyzed (Participants) | 10 | 10
hypoglycemic events
  During Exercise (t=0.5h) | 0 | 2
  During Recovery (t=2.5h) | 1 | 2
  Overnight (t=8h) | 0 | 1

2. Secondary Outcome: Low Blood Glucose Index
Description: A measure of the risk of hypoglycemia. It quantifies the frequency and the extent of low BG readings.
  A LBGI < 2.5 is associated with a low-risk of hypoglycemia, LBGI 2.5-5 is associated with a moderate risk of hypoglycemia, and LBGI > 5 is associated with a high-risk of hypoglycemia.
Time Frame: 26 hours (x2 admissions)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: index score
Arm/Group | Experimental: Heart-Rate Informed SSM+HMM | Control: SSM+HMM
Number analyzed (Participants) | 10 | 10
index score
  During Exercise (t=0.5h) | 0.84 (0.60) | 2.72 (1.61)
  During Recovery (t=2.5h) | 1.81 (1.2) | 1.83 (1.4)
  Overnight (t=8h) | 0.98 (0.41) | 0.49 (0.21)

3. Secondary Outcome: Average Glucose Drop
Description: Average glucose drops at specific time points after the onset of exercise; defined as the difference between plasma glucose at onset of exercise and the glucose values reached at 40 and 60 min post onset of exercise.
Time Frame: 26 hours (2x admissions)
Population: The first two subjects were excluded from the analysis because of protocol violations during the exercise session (the intensity chosen was very high: rating of perceived exertion of 9 out of 10 instead of rating of perceived exertion of 9 out of 20). Results from the 10 remaining subjects are presented.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental: Heart-Rate Informed SSM+HMM | Control: SSM+HMM
Number analyzed (Participants) | 10 | 10
mg/dL
  60 min since exercise onset | -3.4 (12) | -27.7 (10)
  40 min since exercise onset | -5 (10) | -29 (10)

4. Secondary Outcome: Time in Range
Description: Percent time spent within target (70-180 mg/dL) range.
Time Frame: 26 hours (x2 admissions)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of time spent in range
Arm/Group | Experimental: Heart-Rate Informed SSM+HMM | Control: SSM+HMM
Number analyzed (Participants) | 10 | 10
percentage of time spent in range
  Overall | 81 (3.9) | 75 (4.3)
  During Exercise (t=0.5h) | 91 (7.3) | 85 (10.3)
  During Recovery (t=2.5h) | 86 (9.3) | 84 (7.9)
  Overnight (t=8h) | 89 (7.1) | 84 (9.2)

ADVERSE EVENTS:
Groups:
- Experimental: Heart Rate Informed SSM+HMM: Experimental:
  An experimental condition involving an exercise session where the Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) is informed about heart rate
  Heart rate informed SSM+HMM: The Safety Supervision Module + Hyperglycemic Mitigation Module (SSM+HMM) of the Closed Loop is informed about heart rate during exercise. The goal is to demonstrate the feasibility of a modular insulin management system based on continuous glucose monitoring that additionally employs heart rate information to reduce exercise-related hypoglycemic episodes.
Arm/Group | Control: SSM+HMM | Experimental: Heart Rate Informed SSM+HMM
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: SSM+HMM (N=12) | Experimental: Heart Rate Informed SSM+HMM (N=12)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Mild Erythema (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes